CLINICAL TRIAL: NCT03282630
Title: The Effects of Sphenopalatine Ganglion Acupuncture in Patients With Seasonal Allergic Rhinitis: A Randomized Trial
Brief Title: The Effects of Sphenopalatine Ganglion Acupuncture in Patients With Seasonal Allergic Rhinitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TR-acupuncture-2
Record Dates: First submitted 2017-09-06; First posted 2017-09-14 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Patients
Keywords: Acupuncture; Sphenopalatine ganglion; Allergic rhinitis; Randomized Trial
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active acupuncture (Experimental): Procedure/Surgery: active sphenopalatine ganglion acupuncture The acupuncture point was selected in the sphenopalatine ganglion (unilateral side). The acupuncture needle was inserted from the lower border of the zygomatic arch, slightly posterior to the suture protuberance between the zygomatic process and temporal process. The needle was rotated until the participant felt "de-qi" sensations.
  Interventions: Procedure: Sphenopalatine ganglion acupuncture
- sham acupuncture (Sham Comparator): Procedure/Surgery: Sham sphenopalatine ganglion acupuncture The acupuncture point was selected same to the sphenopalatine ganglion. But the needle was inserted at the selected acupuncture site to a depth of only 2-3cm, and the procedure of rotating, twirling and thrusting the needle was repeated, in order to blind the subject to the sham treatment.
  Interventions: Procedure: Sphenopalatine ganglion acupuncture

INTERVENTIONS:
Procedure: Sphenopalatine ganglion acupuncture — * active sphenopalatine ganglion acupuncture The acupuncture point was selected in the sphenopalatine ganglion (unilateral side). The acupuncture needle was inserted from the lower border of the zygomatic arch, slightly posterior to the suture protuberance between the zygomatic process
  * sham sphenopalatine ganglion acupuncture The acupuncture point was selected same to the sphenopalatine ganglion. But the needle was inserted at the selected acupuncture site to a depth of only 2-3cm, and the procedure of rotating, twirling and thrusting the needle was repeated, in order to blind the subject to the sham treatment.

SUMMARY:
Sphenopalatine ganglion (SPG)-acupuncture has been shown to exhibit distinct effects in treatment of nasal inflammatory disease. Investigators aimed to assess the effects of SPG acupuncture in patients with seasonal allergic rhinitis. The randomized, double-blind, controlled clinical trial enrolled participants with seasonal allergic rhinitis. Participants will be randomly assigned to either active SPG-acupuncture group or sham-acupuncture group. All participants will be provided four times of acupuncture in 4 weeks, and then follow-up of 4 week.

Primary trial outcomes are change in symptoms and change in need for medication. The primary outcomes will be measured in baseline, week1, week2, week3, week4, week 6 and week 8. Secondary outcomes include the changes in nasal patency (nasal airway resistance and nasal cavity volume), exhaled nasal nitric oxide.The investigators also evaluate change in neuropeptides (substance P, vasoactive intestinal peptide,neuropeptide Y) and inflammatory cytokines (interleukin(IL)-4, IL-5, IL-8, IL-17a, IL-22, IL-25, interferon-γ, tumor necrosis factor-α, transforming growth factor(TGF)-β1, TGF-β2, TGF-β3,Chemokine, Eotaxin) in nasal secretions as secondary outcomes. The secondary outcomes will be measured in baseline, week1, week4 and week 8.

ELIGIBILITY:
Inclusion Criteria:

* patients with a history of at least 2 years of seasonal allergic rhinitis
* no smoking
* without history of nasal polyps, nasal septum deviation and history of nose surgery) or lung disease (asthma, chronic obstructive pulmonary disease and fibrosis)
* free of upper and lower respiratory tract infections for at least 4 weeks before beginning the study.

Exclusion Criteria:

* had received acupuncture within the last four weeks before the study
* history of diabetes mellitus, autonomic neuropathy, coronary heart disease or hypertension.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2016-01-16 (Actual); Primary Completion 2017-01-16 (Actual); Study Completion 2017-02-20 (Actual)

PRIMARY OUTCOMES:
The change of symptoms | The primary outcomes will be measured in baseline, week1, week2, week3, week4, week 6 and week 8.
  The participants will document the four nasal symptoms (nasal obstruction, rhinorrhea, sneezing, and itching) involved in assigning the total nasal symptom score(TNSS). The symptoms are graded on a four-point scale (0 = no symptoms; 1 = mild symptoms; 2 = moderate symptoms; 3 = severe symptoms). The weekly TNSS will be calculated and compared between the groups.
The change of need for medication | The primary outcomes will be measured in baseline, week1, week2, week3, week4, week 6 and week 8.
  Participants will be asked not to use drugs as much as possible. If drugs are used to relieve symptoms, Medication need will be measured using rescue medication score (RMS), comprising the weekly sum of daily assessments.

SECONDARY OUTCOMES:
The change of nasal patency | The outcomes will be measured in baseline, week1, week4 and week 8.
  Acoustic rhinometry was performed to measure the total nasal cavity volume (cm³) and Rhinomanometer was used to measure the total nasal airway resistance (Pa·cm-³·s-1) .
The change of exhaled nasal nitric oxide | The outcomes will be measured in baseline, week1, week4 and week 8.
  The change of exhaled nasal nitric oxide assessed by nitric oxide analyser. A nitric oxide analyser was used to measure exhaled nasal nitric oxide (nNO). Briefly, NO-free air was aspirated through the nasal cavity at a flow rate of 50 ml/s. The subject exhaled against the air-resistance, resulting in an intraoral pressure to close the velum and prevent mixture of oral and nasal gas. Nasal gas from this circuit was continuously routed in part directly into the analyser for determination of nNO, and the level of nNO(ppb) was calculated from a plateau lasting for at least 3s.
The change of substance P, vasoactive intestinal peptide and neuropeptide Y in nasal secretions | The outcomes will be measured in baseline, week1, week4 and week 8.
  The change of substance P, vasoactive intestinal peptide and neuropeptide Y in nasal secretions were analysed by Enzyme linked immunosorbent assay. Nasal secretions were obtained by inserting a postoperative sinus pack in the nasal cavity (acupuncture side) for five minutes. The quantity of secretions was determined by comparing the weight of the sponges before and after insertion and 2 ml of 0.9% sodium chloride solution was added to each sponge. The sponges were stored at 4°C for two hours and the nasal secretions were recovered from the sponges by centrifugation at 1500 g for 15 minutes at 4°C. The supernatants were separated and stored in aliquots at -20°C until further analysis. The levels of substance P(pg/ml), vasoactive intestinal peptide (ng/ml) and neuropeptide Y (pg/ml) were analysed.
The change of inflammatory cytokines in nasal secretions | The outcomes will be measured in baseline, week1, week4 and week 8.
  The change of inflammatory cytokines (interleukin(IL)-4, IL-5, IL-8, IL-17a, IL-22, IL-25, interferon-γ, tumor necrosis factor-α, transforming growth factor(TGF)-β1, TGF-β2, TGF-β3,Chemokine, Eotaxin) in nasal secretions as secondary outcomes. Nasal secretions were obtained by inserting a postoperative sinus pack in the nasal cavity (acupuncture side) for five minutes. The quantity of secretions was determined by comparing the weight of the sponges before and after insertion and 2 ml of 0.9% sodium chloride solution was added to each sponge. The sponges were stored at 4°C for two hours and the nasal secretions were recovered from the sponges by centrifugation at 1500 g for 15 minutes at 4°C. The supernatants were separated and stored in aliquots at -20°C until further analysis. The levels of inflammatory cytokines (pg/ml) were analysed using the Luminex System.

CONTACTS AND LOCATIONS:
Overall Officials: Chengshuo Wang, Principal Investigator — Beijing Tongren Hospital
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Choi SM, Park JE, Li SS, Jung H, Zi M, Kim TH, Jung S, Kim A, Shin M, Sul JU, Hong Z, Jiping Z, Lee S, Liyun H, Kang K, Baoyan L. A multicenter, randomized, controlled trial testing the effects of acupuncture on allergic rhinitis. Allergy. 2013 Mar;68(3):365-74. doi: 10.1111/all.12053. Epub 2012 Dec 18. PMID 23253122
- [Background] Xue CC, Zhang AL, Zhang CS, DaCosta C, Story DF, Thien FC. Acupuncture for seasonal allergic rhinitis: a randomized controlled trial. Ann Allergy Asthma Immunol. 2015 Oct;115(4):317-324.e1. doi: 10.1016/j.anai.2015.05.017. Epub 2015 Jun 11. PMID 26073163
- [Background] Brinkhaus B, Ortiz M, Witt CM, Roll S, Linde K, Pfab F, Niggemann B, Hummelsberger J, Treszl A, Ring J, Zuberbier T, Wegscheider K, Willich SN. Acupuncture in patients with seasonal allergic rhinitis: a randomized trial. Ann Intern Med. 2013 Feb 19;158(4):225-34. doi: 10.7326/0003-4819-158-4-201302190-00002. PMID 23420231
- [Background] Wang K, Chen L, Wang Y, Wang C, Zhang L. Sphenopalatine Ganglion Acupuncture Improves Nasal Ventilation and Modulates Autonomic Nervous Activity in Healthy Volunteers: A Randomized Controlled Study. Sci Rep. 2016 Jul 18;6:29947. doi: 10.1038/srep29947. PMID 27425415